CLINICAL TRIAL: NCT05533710
Title: Comparative Study Between Bilateral Ultrasound-Guided Erector Spinae Plane Block Versus Bilateral Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative Analgesia After Total Abdominal Hysterectomy
Brief Title: Comparison Between Erector Spinae Plane Block and Transversus Abdominis Plane Block on Postoperative Analgesia After Total Abdominal Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Israa Ihab Abdel Aziz, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ainshamsU FAMSU
Record Dates: First submitted 2022-09-03; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Uterine Diseases
Keywords: ESPB, TAP
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : erector spinae block. (Experimental): patients will receive bilateral ultrasound guided erector spinae block.
  Interventions: Procedure: erector spinae plane block
- Group B : transversus abdominis plane block. (Experimental): patients will receive bilateral ultrasound guided transversus abdominis plane block.
  Interventions: Procedure: transversus abdominis plane block

INTERVENTIONS:
Procedure: erector spinae plane block — Patients will receive ESB. In the lateral decubitus, after skin sterilization, ESP block will be performed at the level of T9
  Arms: Group A : erector spinae block.
Procedure: transversus abdominis plane block — patients will receive TAP block in supine position after skin sterilization, TAP block will be performed between internal oblique and transversus abdominis muscles
  Arms: Group B : transversus abdominis plane block.

SUMMARY:
This study aims to compare the ultrasound-guided bilateral erector spinae block versus the ultrasound-guided bilateral transversus abdominis plane block on postoperative analgesia after total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of Anesthesiologists physical status (ASA) I and II.
2. Female sex.
3. Age between 40 to 60 years old.
4. Scheduled for elective total abdominal hysterectomy surgeries.

Exclusion Criteria:

1. Patient's refusal.
2. Patients who received long-acting opioids preoperatively.
3. Patients with bleeding disorders and coagulopathy.
4. Infection at the injection site.
5. Allergy to local anesthetics.
6. Patients with significant cognitive dysfunction.
7. Patients with diabetic neuropathy.
8. Patients with uncontrolled hypertension or diabetes.
9. Patients with advanced cardiac, respiratory, hepatic or renal disease.
10. Patients with viral hepatitis or HIV.
11. Surgeries which have been complicated or prolonged (more than 150 mins).

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2021-08-28 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperative
  Compare postoperative pain intensity using the total amount of morphine consumption in the first 24 hours after the operation, and the time for first call rescue analgesia
Visual Analog Scale Score | 24 hours postoperative
  Compare postoperative pain intensity using VAS score in the first 24 hours after the operation.The VAS score is a 10-cm line labeled with "worst pain imaginable" on the right border, and "no pain" on the left border (ranging from 0 by indicating no pain to 10 indicating extreme pain).
The time for first call rescue analgesia | 24 hours postoperative
  the time for first call rescue analgesia

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours postoperative
  Measure patient satisfaction by asking the patient if he is satisfied or not "yes or no"
Recognize the adverse effects | 24 hours postoperative
  Recognize the adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: ossama mansour, professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No